CLINICAL TRIAL: NCT06448741
Title: Complete Penile and Testicular Self-amputation: a Very Rare Case
Status: Completed | Type: Observational
Sponsor: Worabe Comprehensive Specialiazed Hospital (Other Government)
Responsible Party: Principal Investigator, Mejudin Kedir Abdella, Urologist, Worabe Comprehensive Specialiazed Hospital
Other Study IDs: Worabe Hospital
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: The Focus of Study is Description of a Very Rare Case

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Replantation of amputated penis — Replantation of the amputated penis done macroscopically, but testicular replantation was not done because of lack of microsurgical access

SUMMARY:
The study is a case report on penile and testicular self-amputation. We didn't assign a drug of intervention. We tried to describe about this rare phenomenon by observation of the presentation and outcome.

DETAILED DESCRIPTION:
We describe a very rare case of bilateral testicular and penile self-amputation by a psychiatric patient who came to our hospital after he amputated his penis and both of his testis. He was operated to replant his severed organs, but because of multiple reasons the replantation failed after 9 days of surgery. This kind of case is very rare, and it is our aim to disseminate the information about the case to physicians for better management in the future.

ELIGIBILITY:
Inclusion Criteria: Patient with Penile and testicular self-amputation -

Exclusion Criteria: Patients with out Penile and testicular self-amputation

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: we studied a single person with unique case
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Replantation | 1 month
  successfully survival of replanted penis

CONTACTS AND LOCATIONS:
Locations (1):
- Worabe Comprehensive Specialized Hospital, Worabe, Ethiopia

IPD SHARING:
Plan to Share IPD: No